CLINICAL TRIAL: NCT00051844
Title: A Double Blind- Randomized, Placebo-controlled Study of Two Doses of Capravirine (AG1549) in Combination With Viracept and Two Nucleoside Reverse Transcriptase Inhibitors in HIV Infected Patients Who Failed an Initial Nonnucleoside Reverse Transcriptase Inhibitor Containing Regimen
Brief Title: Capravirine (AG1549) in Combination With Viracept and Two NRTIs in HIV Infected Patients Who Failed an Initial NNRTI Containing Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4311002
Record Dates: First submitted 2003-01-16; First posted 2003-01-20 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; NNRTI Failure; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — capravirine

INTERVENTIONS:
Drug: Capravirine

SUMMARY:
This is a 48 week study that is intended for HIV Infected persons whose first treatment regimen was with a nonnucleoside reverse transcriptase inhibitor (NNRTI) and who are now failing that regimen. They must be currently on their failing regimen to be eligible.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years old
* HIV RNA level >1000 copies/mL at screening
* CD4 >50 cells/uL at screening
* Patient is currently taking a regimen that includes an NNRTI plus 2 NRTIs for at least 28 days and is currently failing this regimen
* Patient has adequate hematology tests (absolute neutrophil count >1000/uL, Platelets>75,000uL, hemoglobin 9g/L)
* Patient has adequate renal function (serum creatinine of <1.5 upper limit of normal)
* Patient has adequate liver function (AST, ALT, and bilirubin < 2.5 upper limit of normal)

Exclusion Criteria:

* Previous use of protease inhibitors (except if patient has short duration of PI and was switched for tolerability reasons when viral load was <50 copies) This exception does not include Viracept
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2002-08; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
The primary objective was to determine whether the addition of capravirine to a regimen of VIRACEPT and 2 new nucleoside reverse transcriptase inhibitors would provide a higher virologic response rate over 48 weeks
when compared to a 3-drug regimen without capravirine in patients who had experienced virologic failure while on a nonnucleoside reverse transcriptase inhibitor regimen.

SECONDARY OUTCOMES:
The safety and tolerability of 2 doses of capravirine.
The difference between 2 doses of capravirine in terms of tolerability, efficacy, and pharmacokinetics
The relationship of HIV resistance (genotype and phenotype) to virologic response.
The immunologic response as determined by CD4 and CD8 absolute lymphocyte counts
The population pharmacokinetics of capravirine and VIRACEPT
The pharmacokinetics of potential drug-drug interactions.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (28):
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, West Hollywood, California
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Safety Harbor, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Jonesboro, Georgia
  - Pfizer Investigational Site, Tucker, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Stony Brook, New York
  - Pfizer Investigational Site, Huntersville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Akron, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Galveston, Texas
  - Pfizer Investigational Site, Houston, Texas
- France (4):
  - Pfizer Investigational Site, Lyon, Cedex 02
  - Pfizer Investigational Site, Paris, Cedex 10
  - Pfizer Investigational Site, Lyon, Cedex 3
  - Pfizer Investigational Site, Nantes
- Pfizer Investigational Site, Ulm, Bavaria, Germany
- Italy (3):
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
- South Africa (6):
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Johannesburg
  - Pfizer Investigational Site, Pietermaritzburg
  - Pfizer Investigational Site, Port Elizabeth
  - Pfizer Investigational Site, Pretoria North
  - Pfizer Investigational Site, Soweto
- Spain (4):
  - Pfizer Investigational Site, Barakaldo, Bilbao, Vizcaya
  - Pfizer Investigational Site, Bilbao, Vizcaya
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Córdoba